CLINICAL TRIAL: NCT00900913
Title: Effect of Systemic Ropivacaine on Hyperalgesia, Flare Reaction and Peripheral
Brief Title: Effect of Systemic Ropivacaine on Hyperalgesia, Flare Reaction and Peripheral Nerve Excitability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Dr. Konrad Maurer, Institute of Anesthesiology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: StV 24-2008
Record Dates: First submitted 2008-10-21; First posted 2009-05-13 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ropivacaine (Naropin) — intravenous infusion 1 mg/kg bw
  Other Names: Naropin

SUMMARY:
The purpose of this study is to compare the effect of intravenous ropivacaine and lidocaine on the receptive field of primary sensory afferents and their influence on the vascular bed.

*Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

1. Male
2. Age: 18 - 65 years
3. Weight: 50-100kg
4. Height: 155-195cm
5. Signed and dated informed consent
6. Sufficient command of German language

Exclusion criteria:

1. Contraindications to the class of drugs under study
2. Vulnerable subjects (intellectually or mental impaired)
3. Known hypersensitivity to class of drugs or the investigational product
4. Drug abuse
5. Known peripheral neuropathies
6. Diabetes mellitus
7. Chronic alcohol consumption
8. Congestive heart disease
9. Participants of other studies during study period
10. Smoker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Aera of flare reaction (cm2), area of primary and secondary hyperalgesia (cm2) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinical Trial Center, Zurich, Switzerland